CLINICAL TRIAL: NCT03185741
Title: EHR-based Universal Medication Schedule to Improve Adherence to Complex Regimens
Brief Title: Regimen Education and Messaging in Diabetes (REMinD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Emory University (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01NR015444 (NIH)
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UMS Strategy (Experimental): Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions. These materials will be generated within the electronic health record.
  1. Prescription instructions will be adapted to the UMS format to establish four standard time intervals (morning, noon, evening, bedtime) for prescribing and dispensing of medicine. UMS instructions also use simplified text and numeric characters instead of words to detail dose.
  2. Single-page, plain language medication information sheets with important medication-related information following health literacy best practices.
  Interventions: Behavioral: UMS Strategy
- UMS Strategy + SMS Text Messaging (Experimental): In addition to the components from the UMS strategy arm, patients will receive daily text message reminders for 6 months.
  Interventions: Behavioral: UMS Strategy; Behavioral: SMS Text Messaging
- Usual Care (No Intervention): Patients of providers randomized to the usual care arm will receive their standard care

INTERVENTIONS:
Behavioral: UMS Strategy — Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions.
  Arms: UMS Strategy; UMS Strategy + SMS Text Messaging
Behavioral: SMS Text Messaging — Patients will receive daily text message reminders about when to take medicines based on UMS intervals.
  Arms: UMS Strategy + SMS Text Messaging

SUMMARY:
The investigators will leverage increasingly available technologies to impart a Universal Medication Schedule (UMS) in primary care to help patients living with diabetes safely use and adhere to complex drug regimens. The UMS standardizes the prescribing and dispensing of medicine by using health literacy principles and more explicit times to describe when to take medicine (morning, noon, evening, bedtime). This eliminates variability found in the way prescriptions are written by physicians and transcribed by pharmacists onto drug bottle labels. The proposed intervention will standardize prescribing within an electronic health record (EHR) so all medication orders include UMS prescription instructions ('sigs') and patients receive a medication information sheet with their after-visit summaries. Additionally, to help patients remember when to take prescribed medicines we will link unidirectional short message service (SMS) text reminders to the EHR, delivering medication reminders to patients around UMS intervals.

1. Test the effectiveness of the UMS, and UMS + SMS text reminder strategies compared to usual care.
2. Determine if the effects of these UMS strategies vary by patients' literacy skills and language.
3. Using mixed methods, evaluate the fidelity of the two strategies and explore patient, staff, physician, and health system factors influencing the interventions.
4. Assess the costs required to deliver either intervention from a health system perspective.

DETAILED DESCRIPTION:
The investigators will leverage increasingly available technologies to impart a Universal Medication Schedule (UMS) in primary care to help patients living with diabetes safely use and adhere to complex drug regimens. The UMS standardizes the prescribing and dispensing of medicine by using health literacy principles and more explicit times to describe when to take medicine (morning, noon, evening, bedtime). This eliminates variability found in the way prescriptions are written by physicians and transcribed by pharmacists onto drug bottle labels. The proposed intervention will standardize prescribing within an electronic health record (EHR) so all medication orders include UMS prescription instructions ('sigs') and patients receive a medication information sheet with their after-visit summaries. Additionally, to help patients remember when to take prescribed medicines we will link unidirectional short message service (SMS) text reminders to the EHR, delivering medication reminders to patients around UMS intervals.

The investigators will conduct a 3-arm, multi-site trial to test the effectiveness of the UMS, and UMS + SMS text reminder strategies compared to usual care. The investigators will enroll a total of 900 English and Spanish-speaking patients with poorly controlled type 2 diabetes mellitus. Enrolled patients will complete follow-up interviews 3 and 6 months following their baseline interview.

The aims of the investigation are to:

1. Test the effectiveness of the UMS, and UMS + SMS text reminder strategies compared to usual care.
2. Determine if the effects of these UMS strategies vary by patients' literacy skills and language.
3. Using mixed methods, evaluate the fidelity of the two strategies and explore patient, staff, physician, and health system factors influencing the interventions.
4. Assess the costs required to deliver either intervention from a health system perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus diagnosis
2. Most recent hba1c value ≥7.5%.
3. Seek care at participating general internal medicine practices in Chicago or New York City.
4. English or Spanish speaking
5. Take 5 or more prescription drugs for chronic conditions (including 1 study medication)

Exclusion Criteria:

1. Severe uncorrectable vision or hearing impairment
2. Cognitive impairment (≥2 errors on a 6-item dementia screening tool or a chart-documented diagnosis of dementia)
3. Not primarily responsible for administering his/her medications
4. Does not own a cell phone that can receive text messages
5. Not comfortable receiving text messages

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolf, PhD MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- UMS Strategy: Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions. These materials will be generated within the electronic health record.
  1. Prescription instructions will be adapted to the UMS format to establish four standard time intervals (morning, noon, evening, bedtime) for prescribing and dispensing of medicine. UMS instructions also use simplified text and numeric characters instead of words to detail dose.
  2. Single-page, plain language medication information sheets with important medication-related information following health literacy best practices.
  UMS Strategy: Patients of providers randomized to the UMS arm will receive study-related educational tools at their primary care visit to support the understanding, regimen consolidation, and use of prescriptions.
Period: Baseline
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Started | 246 | 272 | 249
Completed | 244 | 267 | 244
Not Completed | 2 | 5 | 5
Not completed — Withdrawal by Subject | 1 | 3 | 2
Not completed — Lost to Follow-up | 1 | 2 | 3
Period: 3Month
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Started | 244 | 267 | 244
Completed | 224 | 242 | 219
Not Completed | 20 | 25 | 25
Not completed — Death | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 5 | 1
Not completed — Lost to Follow-up | 7 | 9 | 8
Not completed — Unavailable for 3Month | 11 | 10 | 11
Not completed — Protocol Violation | 0 | 0 | 3
Period: 6Month
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Started | 235 (Participants who started the 6Month period included those who completed the 3Month period and those who were unavailable for the 3Month period) | 252 (Participants who started the 6Month period included those who completed the 3Month period and those who were unavailable for the 3Month period) | 230 (Participants who started the 6Month period included those who completed the 3Month period and those who were unavailable for the 3Month period)
Completed | 216 | 233 | 211
Not Completed | 19 | 19 | 19
Not completed — Death | 1 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Lost to Follow-up | 16 | 15 | 16

BASELINE CHARACTERISTICS:
Population: Excluded participants with a protocol violation
Groups:
- Total: Total of all reporting groups
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care | Total
Number analyzed (Participants) | 244 | 265 | 241 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.12 (10.69) | 61.82 (10.91) | 60.60 (9.96) | 61.20 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 154 | 141 | 445
  Male | 94 | 111 | 100 | 305
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 7 | 4 | 1 | 12
  Asian | 7 | 9 | 5 | 21
  Black | 105 | 122 | 91 | 318
  Native Hawaiian/Other Pacific Islander | 2 | 0 | 1 | 3
  White | 108 | 120 | 136 | 364
  Other | 1 | 1 | 1 | 3
  More than one race | 14 | 9 | 6 | 29
Recruitment Site [Count of Participants; unit: Participants]
  Northwestern | 118 | 157 | 117 | 392
  Mount Sinai | 126 | 108 | 124 | 358

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence: Pill Count
Description: Adherence will be measured for each prescription medication using an objective pill count of the number of pills within each prescription bottle. The proportion of pills taken over pills prescribed (PT/PP) will be calculated for each medication at baseline and 6Month. Pills taken will be calculated by subtracting the number of pills from the total quantity prescribed. Pills prescribed will be calculated by multiplying the number of pills prescribed each day by the number of days since the medication was filled. A proportion of pills taken over pills prescribed (PT/PP) of 80% or more is considered adherent.
Time Frame: 6 months after baseline
Population: Observations were excluded if: 1.Medications were not in pill form; 2.Participants couldn't provide quantities on their bottles; 3.Missing Fill or Start Dates, 4.Participants started their medications on the same date as their pill count date; 5. Missing medications labels; 6. Participants combined medication bottles and discarded their old bottles; 7. Pills taken > Quantity on bottle; 8. PRN Medications 2 Participants from the UMS Strategy were also excluded due to a Protocol Violation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence (PT/PP =>0.80)
Units Other Than Participants: medications
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Number analyzed (Participants) | 177 | 210 | 182
Number analyzed (medications) | 551 | 725 | 584
Probability of adherence (PT/PP =>0.80) | 0.28 [0.24 to 0.33] | 0.29 [0.25 to 0.34] | 0.30 [0.25 to 0.36]

2. Secondary Outcome: Medication Adherence: 24-hour Recall
Description: Adherence will be measured for each prescription medication using self-report of how many pills and how often each medicine was taken over the last 24 hours. Patients are asked to specify the amount taken (i.e. dose) and when taken (to determine frequency and interval between doses). A patient is considered adherent on a specific medication if they answered all correctly: 1.dose, 2.frequency, 3.interval between doses
Time Frame: 6 months after baseline
Population: Observations were excluded if participants did not complete the 24-hour recall questions.
  2 Participants from the UMS Strategy were also excluded due to a Protocol Violation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of Adherence (Yes)
Units Other Than Participants: medications
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Number analyzed (Participants) | 212 | 229 | 208
Number analyzed (medications) | 1059 | 1192 | 1090
Probability of Adherence (Yes) | 0.72 [0.67 to 0.76] | 0.67 [0.62 to 0.71] | 0.69 [0.64 to 0.73]

3. Secondary Outcome: Medication Adherence: ASK-12
Description: Adherence will be measured by the ASK-12 Adherence Barrier Survey, a subjective assessment of general adherence behaviors and barriers to treatment adherence.
  The ASK-12 is scored by summing the selected responses (with scores ranging from 12 to 60) with higher scores indicating greater barriers to adherence.
Time Frame: 6 months after baseline
Population: Observations were excluded if participants did not complete the ASK12 survey 2 Participants from the UMS Strategy were also excluded due to a Protocol Violation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (12-60)
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Number analyzed (Participants) | 216 | 231 | 208
score on a scale (12-60) | 23.0 [22.23 to 23.82] | 23.89 [23.12 to 24.66] | 23.22 [22.39 to 24.05]

4. Secondary Outcome: Treatment Knowledge
Description: Identification of drug purpose
Time Frame: 6 months after baseline
Population: Observations were excluded if participants did not answer the question. 2 Participants from the UMS Strategy were also excluded due to a Protocol Violation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of Knowledge
Units Other Than Participants: Medications
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
Number analyzed (Participants) | 169 | 180 | 168
Number analyzed (Medications) | 1013 | 1092 | 1007
Probability of Knowledge | 0.73 [0.67 to 0.78] | 0.73 [0.68 to 0.78] | 0.75 [0.70 to 0.80]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | UMS Strategy | UMS Strategy + SMS Text Messaging | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/244 | 2/267 | 4/244
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/267 | 0/244
Other Adverse Events (participants affected / at risk) | 0/244 | 0/267 | 0/244

LIMITATIONS AND CAVEATS:
Due to COVID-19, our recruitment was reduced, approved by the sponsor, from a total sample size of 750 vs. 900 to address new hardships in accessing patients and changes to healthcare delivery. In addition, all interviews were switched to remote vs. in-person data collection. This translated to a remote video interview (Zoom) to capture pill count vs. use of an automated pill counter, and blood pressure could not be collected following the revised protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03185741/Prot_SAP_000.pdf